CLINICAL TRIAL: NCT05480189
Title: Effect of Zoledronic Acid Treatment on Bone-related Events in Breast Cancer Patients With Bone Metastases: a Prospective, Multicenter, Real-world Study
Status: Not yet recruiting | Type: Observational
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Wang Xiaojia, MD, Zhejiang Cancer Hospital
Other Study IDs: IRB-2022-166
Record Dates: First submitted 2022-07-26; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Histologically Confirmed Breast Cancer ,Diagnosis of Bone Metastasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients in breast cancer with bone metastasis: patients in breast cancer with bone metastasis
  Interventions: Other: Non-intervention

INTERVENTIONS:
Other: Non-intervention — Non-intervention,with real world study

SUMMARY:
non-intervention、real world study； Effect of timing and regular treatment of zoledronic acid on the incidence of SREs in breast cancer patients

DETAILED DESCRIPTION:
(1) Main Purpose: To observe the clinical efficacy of zoledronic acid regularly in the prevention of SREs in breast cancer patients with bone metastasis (2) Secondary Objectives:

1. To observe whether zoledronic acid prolonged the time of first SREs in patients with bone metastasis;
2. The clinical efficacy and influencing factors of zoledronic acid in different subgroups were observed by subgroup analysis of population baseline, clinical characteristics (such as different types of breast cancer), past history and complications.
3. To observe the clinical distribution, characteristics, timing and compliance of zoledronic acid administration in Chinese breast cancer patients with first bone metastasis.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years 2. Histologically confirmed breast cancer 3. Initial diagnosis of bone metastasis by MRI or CT and treatment with zoledronic acid 4. Serum creatinine ≤265mol/L or 3.0mg/dl 5. CrCl ≥ 30 ml/min 6. Serum Ca2+ concentration 2.0-3.0 mmonl/L 7.ECOG score ≤2 Voluntary research, informed consent

Exclusion Criteria:

* 1. Pregnant and lactating women 2. Severe liver insufficiency (ALT and/or AST higher than 3 times the upper limit of normal) 3. Patients with osteoarthritis or other bone related diseases need bone targeted therapy 4. Patients with uncontrolled dental problems or planned jaw surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically confirmed breast cancer, Initial diagnosis of bone metastasis
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-08-30 (Estimated); Primary Completion 2023-08-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
SREs | 3 years
  skeletal-related events (SREs) including pathologic fracture, spinal cord compression, hypercalcemia of malignancy, and the need for radiotherapy and/or surgery to bone

SECONDARY OUTCOMES:
time to first on-study SRE | 3 years
  time to first on-study SRE defined as pathologic fracture, radiation or surgery to bone, or spinal cord compression

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojia Wang, MD, Principal Investigator — Zhejiang Cancer Hospital

IPD SHARING:
Plan to Share IPD: Undecided